CLINICAL TRIAL: NCT01261351
Title: Coagulation Activation Markers and Pre Eclampsia : Correlation With Complications
Brief Title: Study of Coagulation Activation Markers and Pre Eclampsia
Acronym: PRESTIGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2008_16/0921; PHRC 2009/1910 (Other Grant/Funding Number: hospital clinical research program, French health ministry); 2009-A00526-51 (Other: ID-RCB number, AFSSAPS)
Record Dates: First submitted 2010-10-26; First posted 2010-12-16 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Pre Eclampsia
Keywords: Pre eclampsia; Endogenous thrombin potential
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Maternal blood and urine
  * cord blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary purpose of the trial is to evaluate coagulation activator markers in patients with pre eclampsia compared to control (normal pregnancy) and to correlate these markers with the severity of the pathology.

DETAILED DESCRIPTION:
100 pre-eclamptic patients will be compared to 200 control patients (100 control matched on gestational age at inclusion and 100 control matched on delivery mode (section).

Blood and urine samples will be collected at PE diagnosis, delivery and post partum.

Two axes will be considered:

1. Thrombography, or kinetic measurement of thrombin generation, by studying the coagulant profile according to Hemker's method in CAT System (Calibrated Automated Thrombogram) and by thromboelastogram in ROTEM technique (delocalized coagulation analyzer), in parallel to specific activation markers (thrombin-antithrombin complex, fibrin monomers).
2. The balance of prostacyclin/thromboxane A2 by using ELISA method for urine samples and genotype-phenotype correlation (Polymorphism of prostacyclin-synthetase's promoter CYP8A1).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* diagnosis of pre eclampsia

Exclusion Criteria:

* multiple pregnancy
* less than 18 year old

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women from two University hospitals in France
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Endogenous thrombin potential | at preeclampsia diagnosis
  comparison of Endogenous thrombin potential between patients with Preclampsia (PE) (at the moment of the diagnosis of PE) compared to control (at the same gestational age)

SECONDARY OUTCOMES:
genotype-phenotype correlation (Polymorphism of prostacyclin-synthetase promoter CYP8A1 | at pre eclampsia diagnosis
In preeclampsia group : correlation between biological markers and severity of the disease | at the diagnosis of preeclampsia
  correlation of endogenous thrombin potential and rotem results with : presence or absence of severe preeclampsia presence or absence of HELLP Syndrome presence or absence of IUGR presence or absence of eclampsia
evolution of endogenous thrombin potential in women with preeclampsia | between the diagnosis of preeclampsia and day 2 of the post partum period
  Study of the evolution of endogenous thrombin potential during the time period of diagnosis of preeclampsia to day 2 of the post partum.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Houfflin Debarge, PHD, Principal Investigator — Universituy Hospital Of Lille, France
Locations (1):
- University Hospital of Lille, Lille, Nord, France